CLINICAL TRIAL: NCT00841074
Title: Effect of Topical Oral Chlorhexidine in Reducing Pneumonia in Nursing Home Residents
Brief Title: Chlorhexidine & Pneumonia in Nursing Home Residents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Catherine J Binkley, PI, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OGMB040944; DE015760
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2016-12

CONDITIONS: Pneumonia; Respiratory Infection
Keywords: Pneumonia; Elderly; Chlorhexidine; Respiratory pathogens
MeSH Terms: conditions — Pneumonia; Respiratory Tract Infections | interventions — Chlorhexidine; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Peridex mouthwash
  Interventions: Drug: chlorhexidine
- 2 (Placebo Comparator): Placebo mouthwash
  Interventions: Drug: Placebo mouthwash

INTERVENTIONS:
Drug: chlorhexidine — 0.12% chlorhexidine mouthwash spray, ~1.3 ml, twice a day.
  Other Names: Peridex
  Arms: 1
Drug: Placebo mouthwash — Placebo mouthwash spray application of ~1.3 ml twice a day.
  Other Names: Peridex mouthwash without chlorhexidine.
  Arms: 2

SUMMARY:
The purpose of this study is determine if topical oral application of a chlorhexidine antimicrobial spray will significantly reduce pneumonia and respiratory infections, and improve oral health compared to a placebo solution in nursing home residents.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be at least 65 years old.
2. Be dependent in 2 or more Activities of Daily Living as noted on the nursing home resident's Minimum Data Set - One must be ADL J- Personal Hygiene.
3. Have natural teeth and/or wear complete or partial dentures.
4. Expected to be a resident in a nursing home for two years.

Exclusion Criteria:

1. Existing pneumonia.
2. History of chlorhexidine reaction or allergy and/or multiple medication or substance allergies.
3. Receiving chlorhexidine oral application at enrollment as prescribed by physician or dentist.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Pneumonia | 12 months

SECONDARY OUTCOMES:
Respiratory pathogens | 12 months
Plaque and Gingival Indices | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J Binkley, DDS, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States